CLINICAL TRIAL: NCT03485040
Title: Defining the Trajectory of Motor Recovery After Stroke
Brief Title: Stroke Motor Rehabilitation and Recovery Study
Acronym: SMaHRT
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Lin, Neurologist, Massachusetts General Hospital
Other Study IDs: 2017P000868
Record Dates: First submitted 2017-12-18; First posted 2018-04-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Stroke, Ischemic
Keywords: Rehabilitation; Neurorehabilitation; Neurotechnology; Neurorecovery; Neurorestoration
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
SMaHRT (Stroke Motor reHabiliation and Recovery sTudy) is a longitudinal study aimed at understanding the natural history of upper extremity motor recovery after ischemic and hemorrhagic stroke.

DETAILED DESCRIPTION:
Participants will be enrolled in the SMaHRT study during their acute stroke hospitalization and will have research visits spanning the post-stroke care continuum at approximately 6 weeks, 3 months, 6 months, one year, two years, and three years after stroke. The study will collect demographics and clinical outcome measures, clinical neuroimages, video and robot-kinematic data and neurophysiology data through TMS and EEG in order to quantify the course of motor recovery. The research visits may be accompanied by a comprehensive clinical visit to the Massachusetts General Hospital Neurorecovery Clinic. The goal is to understand the behavioral, neuroanatomic, and neurophysiologic underpinnings of motor recovery toward developing personalized strategies and neurotechnologies to facilitate neurorehabilitation and enable better recovery for people with stroke.

ELIGIBILITY:
Inclusion Criteria

* Age 18 - 90
* Upper extremity motor weakness after ischemic and/or hemorrhagic stroke as defined by a score of >=1 on NIH Stroke Scale Arm Motor Drift Questions 5A or 5B
* Ability to follow simple commands in English
* Score of zero or 1 on the NIH Stroke Scale Level of Consciousness Questions 1a and 1b and a score of zero on the NIH Stroke Scale Level of Consciousness Question 1c.
* Stable medical status as determined by primary care team
* Inpatient on the MGH stroke neurology service

Exclusion Criteria

* Prior history of developmental, neurologic, or major psychiatric disorder resulting in functional disability
* Prior history of visual or auditory disorders limiting ability to participate in testing
* Evidence of an uncontrolled seizure disorder
* Patients for whom EEG leads are contraindicated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to the Massachusetts General Hospital with upper extremity motor weakness after ischemic and/or hemorrhagic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-06-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Arm Motor Assessment | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This test provides information about level of upper extremity motor impairment after stroke. The test includes a series of different movements that allow for the assessment of functional movement capacity and quality. The scale is used to track change in upper extremity motor impairment over the course of one year post stroke.

OTHER OUTCOMES:
Barthel Index | Time 1: During acute hospitalization; Time 2: ~ 6 weeks after stroke date; Time 3: ~ 90 days after stroke date; Time 4: ~ 180 days after stroke date; Time 5: ~ 1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This test provides information about independence/dependence in performing activities of daily living (ADLs). The test includes a series of questions which can be asked of the patient, a care giver, or member of the medical team. The scale is used to track independence with ADLs over the course of one year post stroke.
Pre-Morbid Modified Rankin Score | Time 1: During acute hospitalization; Time 2: N/A; Time 3: N/A; Time 4: N/A; Time 5: N/A Time 6: N/A; Time 7: N/A
  This scale is used to measure degree of disability based on functional status. The scale involves a series of questions asked to determine the degree of disability prior to stroke. A lower score indicates less disability. Scores range from zero to 6 with zero representing no disability and 6 representing death. The scale increments by units of 1.
Current Modified Rankin Score | Time 1: During acute hospitalization; Time 2: ~ 6 weeks after stroke date; Time 3: ~ 90 days after stroke date; Time 4: ~ 180 days after stroke date; Time 5: ~ 1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This scale is used to measure degree of disability based on functional status. The scale involves a series of questions asked to determine the degree of disability a participant is experiencing at the current timepoint. The scale is used to track a participant's degree of disability over the course of one year post stroke.
Patient Health Questionnaire 2 and 9 | Time 1: During acute hospitalization; Time 2: ~ 6 weeks after stroke date; Time 3: ~ 90 days after stroke date; Time 4: ~180 days after stroke date; Time 5: ~ 1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This questionnaire is used to screen, diagnose, and monitor post stroke depression. The questionnaire includes a series of questions which allow a participant to self-report how often he/she has been experiencing symptoms of depression. The questionnaire is used to track mental health over the course of one year post stroke.
Stoke Impact Scale 16 | Time 1: N/A; Time 2: ~ 6 weeks after stroke date; Time 3: ~90 days after stroke date; Time 4: ~ 180 days after stroke date; Time 5: ~ 1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This questionnaire is used to monitor a participant's self-reported reflection of how difficult it is to perform his/her activities of daily living. The questionnaire includes a series of questions that the participant is asked to rate in terms of level of difficulty. The scale is used to track participant impression over the course of the participant's outpatient treatment.
National Institute of Health Stroke Scale | Time 1: During acute hospitalization; Time 2: ~ 6 weeks after stroke date; Time 3: ~ 90 days after stroke date; Time 4: ~ 180 days after stroke date; Time 5: ~ 1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This test provides information about overall stroke severity. The test includes a series of different questions which allow for the assessment of level of consciousness, vision, facial, arm, and leg motor weakness, sensation, coordination, and language expression and reception. The scale is used to track nervous system recovery over the course of one year post stroke.
Dynamometer | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This activity is used to measure a participant's grip strength. The test requires the participant to squeeze an instrument called a dynamometer with each hand three times. The activity is used to track change in grip strength bilaterally over the course of one year post stroke.
Box and Blocks | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This activity is used to assess a participant's coordination, dexterity, and gross upper extremity motor function. The test requires the participant to move blocks from one side of a box to the other with his/her unaffected hand and then his/her affected hand, with the goal of moving as many blocks as possible in one minute. The activity is used to track progress of both fine and gross upper extremity motor function over the course of one year post stroke.
Nine Hole Peg Test | Time Frame: Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This activity is used to assess a participant's upper extremity coordination and fine motor skills. The test requires the participant to place nine pegs into nine holes, one at a time, and then to remove each peg one at a time with his/her unaffected hand and then his/her affected hand, with the goal of performing the task in the shortest amount of time possible. The activity is used to track progress in both coordination and fine motor function over the course of one year post stroke.
Gait Velocity Test | Time Frame: Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This activity is used to assess a participant's level of ambulation from house hold ambulator to limited community ambulator to community ambulator. The test requires the participant to walk 10 meters twice. The middle six meters are timed to determine a participant's gait velocity. The test is used to track ambulation status over the course of one year post stroke.
Timed Up and Go | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This activity is used to assess a participant's fall risk. The test requires the participant to sit in a chair, walk 3 meters, turn around, walk 3 meters, and sit back down in the chair. The test is used to track fall risk over the course of one year post stroke.
Overall Impressions of Level of Recovery and Level of Disability | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This test is used to assess a participant's impression of how his/her arm weakness affects his/her everyday life, and impression of overall recovery following stroke. The participant is asked both to rate arm weakness and overall recovery on a scale from 0 to 10, with 10 being the worst weakness, no recovery and zero being complete strength and full recovery. The test is used to track participant impression of weakness and recovery over the course of one year post stroke.
PROMIS Scale | Time 1: N/A; Time 2: ~ 6 weeks after stroke date; Time 3: ~ 90 days after stroke date; Time 4: ~ 180 days after stroke date; Time 5: ~ 1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This questionnaire is used to assess a participant's impression of his/her global physical health and global mental health. The participant is asked a series of questions about his/her health and given rating scales for each question. The test is used to track participant impression of physical and mental health over the course of the participant's outpatient treatment.
Shoulder Abduction / Finger Extension (SAFE) | Time 1: During acute hospitalization; Time 2: ~ 6 weeks after stroke date; Time 3: ~ 90 days after stroke date; Time 4: ~ 180 days after stroke date; Time 5: ~ 1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This test is used to assess MRC (Medical Research Council) muscle strength grading of shoulder abduction and finger extension.
Modified Ashworth Scale (MAS) | Time 1: N/A; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This test is used to assess spasticity at different joints of the upper extremity. The greatest MAS score at the shoulder, elbow, wrist, fingers will be taken.
Edinburgh Handedness Inventory | Time 1: During acute hospitalization; Time 2: N/A; Time 3: N/A; Time 4: N/A; Time 5: N/A; Time 6: N/A; Time 7: N/A
  This screener is used to identify the handedness of participants prior to stroke by asking them which hand they typically use to complete activities of daily living, such as writing, throwing a ball, cutting paper with scissors, brushing teeth, and eating with a spoon. Participants can answer if they would use strictly their right hand, right more than left, both equally, left more than right, or strictly their left hand. Participants are then categorized as left-handed, ambidextrous, or right-handed.
Rehabilitation Therapy | Time 1: N/A; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This measure helps quantify how much therapy a participant receives once s/he is discharged after acute stroke hospitalization. It asks participants which modalities of therapies they have received, such as occupational, physical, or speech, and the setting it took place (e.g., home, outpatient, inpatient). Furthermore, patients are asked if they met with a psychologist or psychiatrist since the previous timepoint.
Functional Ambulation Category (FAC) | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date Time 6: N/A; Time 7: N/A
  This test is used to evaluate how much support participants need while ambulating. Outcomes range from non-ambulatory to walking on unlevel ground and stairs independently.
Montreal Cognitive Assessment (MoCA) | Time 1: During acute hospitalization; Time 2: ~ 6 weeks after stroke date; Time 3: ~ 90 days after stroke date; Time 4: ~ 180 days after stroke date; Time 5: ~1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This test is used to assess cognitive dysfunction by testing multiple different cognitive domains including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
Cognitive Linguistic Quick Test (CLQT) | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date; Time 6: N/A; Time 7: N/A
  This assessment measures the status of cognitive-linguistic functioning in five cognitive domains (Attention, Memory, Executive Functions, Language, and Visuospatial Skills).
Quick Aphasia Battery (QAB) | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date; Time 6: N/A; Time 7: N/A
  This assessment provides a reliable and multidimensional assessment of language function. Eight summary measures are derived, including word and sentence comprehension, word finding, grammatical construction, speech motor programming, repetition, and reading.
Social Determinants of Health | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date; Time 6: N/A; Time 7: N/A
  This survey is used to better understand the socioeconomic status and demographics of participants in the study.
User Participation | Time 1: N/A; Time 2: N/A; Time 3: N/A; Time 4: approx. N/A; Time 5: approx. 1 year after stroke date; Time 6: N/A; Time 7: N/A
  This questionnaire is used to quantify participants' participation in daily life activities, the amount of time spent on them, limitations they may experience, and their satisfaction with such.
4AT - Rapid Clinical Test for Delirium Detection | Time 1: During acute hospitalization; Time 2: approx. 6 weeks after stroke date; Time 3: approx. 90 days after stroke date; Time 4: approx. 180 days after stroke date; Time 5: approx. 1 year after stroke date; Time 6: N/A; Time 7: N/A
  This screening instrument is used to determine if a participant displays signs of delirium.
Sleep Condition Indicator | Time 1: N/A; Time 2: ~ 6 weeks after stroke date; Time 3: ~90 days after stroke date; Time 4: ~ 180 days after stroke date; Time 5: ~ 1 year after stroke date Time 6: ~ 2 years after stroke date; Time 7: ~ 3 years after stroke
  This questionnaire is used to evaluate sleep by asking participants about concerns going to sleep, remaining asleep, quality of sleep, and how it affects daytime quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: David J Lin, MD, Principal Investigator — Neurologist
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kline DK, Lin DJ, Cloutier A, Sloane K, Parlman K, Ranford J, Picard-Fraser M, Fox AB, Hochberg LR, Kimberley TJ. Arm Motor Recovery After Ischemic Stroke: A Focus on Clinically Distinct Trajectory Groups. J Neurol Phys Ther. 2021 Apr 1;45(2):70-78. doi: 10.1097/NPT.0000000000000350. PMID 33707402
- [Background] Lin DJ, Erler KS, Snider SB, Bonkhoff AK, DiCarlo JA, Lam N, Ranford J, Parlman K, Cohen A, Freeburn J, Finklestein SP, Schwamm LH, Hochberg LR, Cramer SC. Cognitive Demands Influence Upper Extremity Motor Performance During Recovery From Acute Stroke. Neurology. 2021 May 25;96(21):e2576-e2586. doi: 10.1212/WNL.0000000000011992. Epub 2021 Apr 15. PMID 33858997
- [Background] Kuo YL, Lin DJ, Vora I, DiCarlo JA, Edwards DJ, Kimberley TJ. Transcranial magnetic stimulation to assess motor neurophysiology after acute stroke in the United States: Feasibility, lessons learned, and values for future research. Brain Stimul. 2022 Jan-Feb;15(1):179-181. doi: 10.1016/j.brs.2021.12.001. Epub 2021 Dec 7. No abstract available. PMID 34890840